CLINICAL TRIAL: NCT06915519
Title: Predictive Value Of Muscle Tone Loss And Perfusion Index In The Success Of Supraclavicular Brachial Plexus Block: A Pilot Study
Brief Title: Predictive Value Of Muscle Tone And Perfusion Index In Supraclavicular Block Success.
Acronym: PREVAM
Status: Completed | Type: Observational
Sponsor: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Gloria Fabiola Alvarez-Orenday, Anesthesiologist, Hospital Central "Dr. Ignacio Morones Prieto"
Other Study IDs: CONBIOETICA-24-C1-20160427
Record Dates: First submitted 2025-03-18; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Regional Anesthesia Success; Orthopedic Surgery
Keywords: supraclavicular block; regional anesthesia; perfusion index; motor strength
MeSH Terms: interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: measure motor strength and perfusion index — measurements of the motor strength and perfusion index in the blocked hand to predict the successfulness of the supraclavicular block at 0, 5, 10 and 15 min post blockage.

SUMMARY:
The goal of this observational study is to define the usefulness of a new device to predict the supraclavicular block successfulness in the patients scheduled to orthopedic surgery. The main question it aims to answer is:

¿The combination between a flexometer and perfusion index is capable to predict the successfulness of a supraclavicular block in the first 15 min?

Participants will be anesthetized by residents or anesthesiologist with regional anesthesia training and then connected to a flexometer to measure the motor blockade and a pulse oximeter to measure the perfusion index related to sympathetic blockage at 0, 5, 10 and 15 min .

DETAILED DESCRIPTION:
Prospective observational pilot study conducted at "Dr. Ignacio Morones Prieto" Central Hospital, Mexico, involving 33 patients (ASA 1, 2, 3) requiring surgery on the distal third of the upper limb with ultrasound-guided SCPB. The motor block was assessed with a conductive ink flexion sensor, and the sympathetic block was evaluated with perfusion index via pulse oximeter at 3, 5, 10, and 15 minutes. Block success was defined as a Numerical Rating Scale (NRS) for pain <2 during surgical stimulation. Statistical comparisons were made between successful and unsuccessful blocks, with ROC curve analysis identifying optimal cutoff points for predictive variables.

ELIGIBILITY:
Inclusion Criteria:

* patients with 18 years and older.
* ASA 1, 2, and 3.
* patients who required surgical intervention in the distal two-thirds of an upper limb and warranted the application of an ultrasound-guided supraclavicular brachial plexus block.

Exclusion Criteria:

* infection at the puncture site
* allergy to local anesthetics
* diagnosis of coagulopathy
* restrictive pulmonary pathology
* diaphragmatic pathology
* dependence on supplemental oxygen
* brachial plexus radiculopathy
* uncontrolled type 2 diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled to orthopedic surgery of the upper limb in the Hospital General "Dr. Ignacio Morones Prieto" in San Luis Potosi, Mexico.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
measurement of motor strength with the flexometer in the blocked hand at 0, 5, 10, 15 minutes post blockage | Periprocedural
  the patient will be asked to move the third finger of the blocked hand which will be connected to the flexometer to measure the motor strength at 0, 5, 10 and 15 minutes and correlate with the successfulness of the block.
measurement of sympathetic block with perfusion index in the blocked hand | Periprocedural
  measurement of the perfusion index in the blocked hand at 0, 5, 10 and 15 minutes post blockage and correlate with the sympathetic block and successfulness of the supraclavicular block.

SECONDARY OUTCOMES:
success of supraclavicular block | Periprocedural
  measure the success of the block defined as Numeric Scale Rate (NRS from 0 to 10) less 2 and absence to change the anesthetic technique during the surgery. Less NRS is correlated with successfulness of the blockage.

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Govea-Hernandez, Anesthesiologist, Study Director — anesthesia department; Mauricio Guerra-Hernandez, Medical Doctor, Study Chair — Anesthesiology Departmen; Venance Basil-Kway, Medical Doctor, Study Director — Clinical Investigation Department
Locations (1):
- Hospital General "Dr. Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
at the moment, the patients data are confidential, so, we haven't decide to share with other investigators. only data used in the results will be available.

REFERENCES:
- [Background] Roy M, Nadeau MJ, Cote D, Levesque S, Dion N, Nicole PC, Turgeon AF. Comparison of a single- or double-injection technique for ultrasound-guided supraclavicular block: a prospective, randomized, blinded controlled study. Reg Anesth Pain Med. 2012 Jan-Feb;37(1):55-9. doi: 10.1097/AAP.0b013e3182367b97. PMID 22030724
- [Background] Perlas A, Lobo G, Lo N, Brull R, Chan VW, Karkhanis R. Ultrasound-guided supraclavicular block: outcome of 510 consecutive cases. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):171-6. doi: 10.1097/AAP.0b013e31819a3f81. PMID 19282715
- [Background] Vásquez, M., Jiménez, A., Aguirre, O., Gonzalez, M., y Ríos, A. (2012). Bilateral ultrasound-guided supraclavicular block. Revista colombiana de anestesiología, 40(4), 304-308.
- [Background] Mian A, Chaudhry I, Huang R, Rizk E, Tubbs RS, Loukas M. Brachial plexus anesthesia: A review of the relevant anatomy, complications, and anatomical variations. Clin Anat. 2014 Mar;27(2):210-21. doi: 10.1002/ca.22254. Epub 2013 Aug 20. PMID 23959836
- [Background] Dzul-Martín, C., y Torres-Anaya, C. (2016). Actualidades en el bloqueo de plexo braquial. Revista mexicana de anestesiología, 39(1), 272-275.